CLINICAL TRIAL: NCT04747639
Title: Double-blind, Randomized, Controlled, Four Treatment Four Period Cross-over Trial on Glycemic Response, Excretion of Gluconate and Tolerability of Two Doses of Low Sugar Apple Juice
Brief Title: Glycemic Response to Two Doses of Low Sugar Apple Juice
Acronym: HB-RCT2-2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Center Kiel GmbH (Other)
Collaborators: Nofima (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HB-RCT2-2015
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-02

CONDITIONS: Prediabetes
Keywords: glycemic response, enzymatic conversion, gluconate
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: a double-blind randomised controlled cross-over trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The test products (verum and control) are similar in flavour, color, texture, appearance and identical in packaging to ensure the double-blind, controlled design of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- verum 500 (Active Comparator): 500 ml low sugar apple juice manufactured from conventional apple juice via a series of enzymatic reactions that end up in a final content of free glucose less than 0,5 g/l.
  Interventions: Other: 500 ml glucose-depleted apple juice
- control 500 (Placebo Comparator): 500 ml conventional apple juice produced by a general apple juice production process (free glucose 17g/l)
  Interventions: Other: 500 ml conventional apple juice
- verum 250 (Active Comparator): 250 ml low sugar apple juice manufactured from conventional apple juice via a series of enzymatic reactions that end up in a final content of free glucose less than 0,5 g/l.
  Interventions: Other: 250 ml glucose-depleted apple juice
- control 250 (Placebo Comparator): 250 ml conventional apple juice produced by a general apple juice production process (free glucose 17g/l)
  Interventions: Other: 250 ml conventional apple juice

INTERVENTIONS:
Other: 500 ml glucose-depleted apple juice
  Arms: verum 500
Other: 500 ml conventional apple juice
  Arms: control 500
Other: 250 ml glucose-depleted apple juice
  Arms: verum 250
Other: 250 ml conventional apple juice
  Arms: control 250

SUMMARY:
Single center, double-blind, randomized controlled cross-over trial with four treatments and four time points.

The study has three primary objectives. The first primary objective is to confirm the reduction of postprandial glycemic and insulinemic response after consumption of 500 ml glucose-free apple juice compared to 500 ml untreated apple juice as could be shown in a previous study

DETAILED DESCRIPTION:
Single center, double-blind, randomized controlled cross-over trial with four treatments and four time points.

The study has three primary objectives. The first primary objective is to confirm the in a previous study shown reduction of postprandial glycemic and insulinemic response after consumption of 500 ml glucose-free apple juice compared to 500 ml untreated apple juice.

The second primary objective is to show the reduction of postprandial glycemic response after consumption of 250 ml glucose-free apple juice compared to 250 ml untreated apple juice.

The third primary objective is to show the reduction of insulinemic response after consumption of 250 ml glucose-free apple juice compared to 250 ml untreated apple juice.

Secondary objectives include safety aspects, specifically the occurrence of diarrhoea in all four treatment groups, differences between treatment groups on the Bristol Stool Forms Scale, gastro-intestinal symptoms and laboratory parameters. In addition, gluconate excretion and excreted portion of ingested gluconate are of interest as well as faecal pH.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥ 18y
2. Impaired fasting glucose (IFG)
3. Written informed consent
4. Consent to collect stools and urine four times for three days

Exclusion Criteria:

1. Subjects currently enrolled in another clinical study
2. Subjects having finished another clinical study within the last 4 weeks before inclusion.
3. Subjects having participated in the study HB-RCT1-2015
4. Hypersensitivity, allergy or idiosyncratic reaction to apple, apple juice or other apple containing food
5. Acute or chronic infections
6. Renal insufficiency
7. Gastrointestinal illness
8. No stools of type 5-7 of Bristol Stool Form Scale within the last week before inclusion
9. History of gastrointestinal surgery
10. Known fructose intolerance
11. Overt diabetes mellitus
12. Endocrine disorders
13. Any disease or condition which might compromise significantly the hematopoietic, renal, endocrine, pulmonary, hepatic, cardiovascular, immunological, central nervous, dermatological or any other body system with the exception of the conditions defined by the inclusion criteria
14. History of hepatitis B and C
15. History of HIV infection
16. History of coagulation disorders or pharmaceutical anti-coagulation (with the exception of acetylsalicylic acid)
17. Regular medical treatment including OTC, which may have impact on the study aims (e.g. gluconic acid-containing OTCs, antidiabetic drugs, laxatives etc.)
18. Major cognitive or psychiatric disorders
19. Subjects who are scheduled to undergo hospitalization during the study period
20. Eating disorders (e.g. anorexia, bulimia) or special diets (e.g. vegan, vegetarian)
21. Present drug abuse or alcoholism
22. Legal incapacity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
iAUC glucose 500 | 120 min after ingestion
  Incremental AUC (iAUC120) of blood glucose levels (according to FAO/WHO) after 500 ml juice
iAUC insulin 500 | 120 min after ingestion
  iAUC insulin 500
iAUC glucose 250 | 120 min after ingestion
  Incremental AUC (iAUC120) of blood glucose levels (according to FAO/WHO) after 250 ml juice
iAUC insulin 250 | 120 min after ingestion
  iAUC insulin 250

SECONDARY OUTCOMES:
diarrhea | before and 60 and 120 minutes after ingestion with respect to the last 2 hours
  Occurrence of diarrhoea as assessed by stool frequency and Bristol Stool Forms Scale (Lewis, 1997) (3 or more loose or liquid stools per day, definition according to the WHO)
gastro-intestinal symptoms | before and 60 and 120 minutes after ingestion with respect to the last 2 hours
  Assessed by completing questionnaires on gastrointestinal symptoms (GSRS; Svedlund 1988; Dimenäs 1995; Revicki 1998)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Laue, Dr. (MD), Principal Investigator — CRC Clinical Research Center Kiel
Locations (1):
- CRC Clinical Research Center Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No